CLINICAL TRIAL: NCT03921515
Title: Skin Immunity Sample Collection Involving Blisters and Biopsies
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study closed by PI, no enrollment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190084; 19-I-0084
Record Dates: First submitted 2019-04-18; First posted 2019-04-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hyper-Immunoglobulin E. Syndrome (HEIS); Chronic Granulomatous Disease (CGD)
Keywords: Hyper-Immunuglobulin E.Syndrome; Chronic Granulomatous Disease; Tumor Necrosis Factor Alpha; Staphylococcus Aureus
MeSH Terms: conditions — Granulomatous Disease, Chronic; Staphylococcal Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Other): Blister Induction
  Interventions: Other: Blister induction
- 2 (Other): Skin Biopsies
  Interventions: Other: Skin Biopsies

INTERVENTIONS:
Other: Blister induction — Blister induction involves creating 8 blisters on the forearm and removing the tops of the blisters for primary cell culture derivation. After blister induction, subjects may have an optional overnight admission to assess cell infiltration in response to autologous serum and/or sterile saline solution.
  Arms: 1
Other: Skin Biopsies — The skin biopsies will involve up to 4 biopsies: 2 initial punch biopsies 2 mm in diameter, followed by a punch biopsy 3 (plus or minus 1) and 7 (plus or minus 2) days later using a 3 mm punch to encompass the initial biopsy sites, capturing the tissue at 3 and 7 days of healing.
  Arms: 2

SUMMARY:
Background:

The way the body heals and protects itself from getting sick is called the immune response. Some people with weak immune systems get sick often or get rashes and skin infections. Researchers want to find out how the immune system and skin problems are related so they can help these people.

Objective:

To learn about how immune response and skin healing are related to each other.

Eligibility:

People ages 18-65 with hyper IgE syndrome or Job syndrome or people ages 7-65 with chronic granulomatous disease. Healthy volunteers ages 18 65 are also needed.

Design:

Participants will be screened with:

Medical history

Physical exam

Possible urine tests

Participants will have 1 to 3 visits within about a week. Visits will include the following:

Participants will have a wells device strapped to the inside of the forearm. It will suction the skin and pull the top layer away to form 8 blisters. The skin over the blisters and the liquid inside will be collected.

Participants will have up to 4 skin biopsies. A sharp tool will remove a small plug of skin from the forearm.

Participants may have blood and urine tests.

The skin on participants skin will be rubbed with a cotton swab.

Some participants will have an overnight visit. They will have the blister device placed back on the arm. The wells will be lined up over the blister wounds. The wells will be filled with either saline or the participant s blood serum. The device will be covered and left on the arm for up to 24 hours. Doctors will periodically remove some liquid from the wells.

DETAILED DESCRIPTION:
The incidence of community-associated (CA) staphylococcal infections, especially those caused by methicillin-resistant Staphylococcus aureus (MRSA), has increased in recent years. Skin and soft tissues are the primary sites for these infections. Although many patients without apparent underlying immune dysfunction suffer from recurrent and persistent skin infections with S.aureus, patients with conditions such as hyper immunoglobulin E syndrome (HIES, or Job s syndrome) and chronic granulomatous disease (CGD) are disproportionately affected. Although underlying host molecular defects responsible for some of these predisposing conditions have been uncovered in recent years, the skin immune response to S. aureus infections has not been elucidated in either healthy volunteers or susceptible populations. We hypothesize that the local skin response determines susceptibility to S. aureus skin infection.

In this sample collection protocol, we will perform exploratory evaluations of anti-staphylococcal immune responses in healthy volunteers, subjects with HIES, and subjects with CGD. Following screening and baseline procedures, including blood draw and skin swab, subjects will have the option to undergo blister induction, where a suction device will be used to induce skin blisters on the forearm. The tops of the blisters and blister fluid will be collected for research testing and storage for future research. An optional overnight inpatient stay may be performed to collect additional cellular infiltrates in response to autologous serum and/or sterile saline. Subjects may also have up to 4 skin punch biopsies from the forearm over the course of a week to capture wound healing progress and identify involved genes. All research procedures will be performed at the National Institutes of Health Clinical Center (NIH CC).

The primary objective of this research is to perform ex vivo assessment of wound healing pathways using a skin blister model and skin biopsies to obtain keratinocyte cultures and evaluate skin immune responses. We will use three experimental approaches: 1) ex vivo evaluation of anti-microbial responses and tissue remodeling through derivation of keratinocyte cultures from skin blisters and biopsies, 2) in vivo and ex vivo assessment of cellular response after blister induction using overnight exposure to autologous serum and/or sterile saline, and 3) evaluation of in vivo responses to skin biopsies. We anticipate that the research will provide critical new information on the human skin immune and remodeling responses and will have direct relevance for the development of vaccines, diagnostics, and therapeutics.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Meets one of the following:

     1. has documentation of HIES or CGD (patient populations); or
     2. does not have clinically apparent evidence of an immune defect or history of invasive or recurrent S. aureus infections (healthy volunteers).
  2. Between the following age limits (inclusive):

     1. 18 and 65 years old for healthy volunteers;
     2. 7 and 65 years old for patients with CGD;
     3. 18 and 65 years old for patients with HIES.
  3. Willing to allow storage of blood, RNA, bacterial and fungal cultures, and other tissue samples for future research.
  4. Able to provide informed consent.

EXCLUSION CRITERIA:

The following exclusion criteria apply to all subjects:

1. For individuals undergoing blister or skin biopsy procedures, history of keloid formation.
2. Current or prior (within 3 months) anticoagulant or anti-platelet therapy (other than aspirin or non-steroidal anti-inflammatory drugs [NSAIDs]).
3. Current or prior (within 3 months) use of immunomodulatory drugs (e.g., chemotherapy, steroids), except if approved by the principal investigator.
4. Pregnancy.
5. Any condition that, in the opinion of the investigator, contraindicates participation in the study.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Tumor necrosis factor alpha (TNFa) production by keratinocytes from patients with HIES versus healthy volunteers | Throughout study
  Evaluate epithelial cell responses to cutaneous wounds and infections of keratinocytes and other cutaneous epithelial cells in patients with HIES or CGD and healthy volunteers.
T-cell infiltration as percent of total cell infiltration in patients with CGD versus healthy volunteers. | Throughout study
  Identify cellular mediators that contribute to the inflammatory processthrough evaluation of infiltrating cell types.
Fold induction in genes related to wound healing. | Throughout study
  Determine whether there are abnormalities in specific tissue repair pathways, such as epithelial to mesenchymal transition (EMT).

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Myles, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Klevens RM, Morrison MA, Nadle J, Petit S, Gershman K, Ray S, Harrison LH, Lynfield R, Dumyati G, Townes JM, Craig AS, Zell ER, Fosheim GE, McDougal LK, Carey RB, Fridkin SK; Active Bacterial Core surveillance (ABCs) MRSA Investigators. Invasive methicillin-resistant Staphylococcus aureus infections in the United States. JAMA. 2007 Oct 17;298(15):1763-71. doi: 10.1001/jama.298.15.1763. PMID 17940231
- [Background] Naimi TS, LeDell KH, Como-Sabetti K, Borchardt SM, Boxrud DJ, Etienne J, Johnson SK, Vandenesch F, Fridkin S, O'Boyle C, Danila RN, Lynfield R. Comparison of community- and health care-associated methicillin-resistant Staphylococcus aureus infection. JAMA. 2003 Dec 10;290(22):2976-84. doi: 10.1001/jama.290.22.2976. PMID 14665659
- [Background] Myles IA, Datta SK. Staphylococcus aureus: an introduction. Semin Immunopathol. 2012 Mar;34(2):181-4. doi: 10.1007/s00281-011-0301-9. Epub 2012 Jan 27. No abstract available. PMID 22282052
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-I-0084.html